CLINICAL TRIAL: NCT06584305
Title: Artificial Intelligence Screening for Body Dysmorphic Disorder in Aesthetic Surgery: Improving Patient Safety and Outcomes
Brief Title: AI Screening for BDD in Aesthetic Surgery: Enhancing Safety and Outcomes
Acronym: AI
Status: Completed | Type: Observational
Sponsor: Bukret Plastic Surgery (Other)
Responsible Party: Sponsor
Other Study IDs: BukretAI-BDD2024
Record Dates: First submitted 2024-08-30; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Body Dysmorphic Disorder
Keywords: Body Dysmorphic Disorder; Artificial Intelligence; BDD Screening; Aesthetic Surgery; Cosmetic Surgery; AI-based Risk Assessment; Patient Safety; Psychological Screening; Plastic Surgery; Mental Health in Surgery; prevention
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AI-Screened Cosmetic Surgery Patients: This cohort consists of patients aged 18 years or older who are undergoing elective cosmetic surgery. All participants in this group have undergone an AI-powered Body Dysmorphic Disorder (BDD) screening, which includes the completion of the Body Dysmorphic Disorder Questionnaire (BDDQ) and additional psychological evaluations. The AI system provides a risk assessment for BDD, guiding the surgical decision-making process and identifying patients who may require psychological intervention before proceeding with surgery.
  Interventions: Procedure: AI-Powered Body Dysmorphic Disorder Screening Procedure

INTERVENTIONS:
Procedure: AI-Powered Body Dysmorphic Disorder Screening Procedure — The AI-Powered Body Dysmorphic Disorder Screening Procedure involves using an AI tool to evaluate patients for Body Dysmorphic Disorder (BDD) before undergoing elective cosmetic surgery. The screening integrates the Body Dysmorphic Disorder Questionnaire (BDDQ) with additional psychological assessments. The AI system processes the collected data to produce a risk score, guiding surgeons in making informed decisions about the need for psychological evaluation or intervention, and determining the suitability of patients for surgery.

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of an AI-powered screening tool for Body Dysmorphic Disorder (BDD) among patients seeking aesthetic surgery. The study aims to determine if the AI system can effectively identify patients at risk for BDD and assess the impact of early psychological intervention on surgical decision-making and outcomes. Participants will complete a comprehensive AI-based risk assessment, which includes the Body Dysmorphic Disorder Questionnaire (BDDQ). The study will track the correlation between BDD, age, stress levels, and gender to better understand the prevalence and implications of BDD in cosmetic surgery.

DETAILED DESCRIPTION:
This observational study evaluates an AI-powered screening tool for Body Dysmorphic Disorder (BDD) in patients seeking elective aesthetic surgery. The study is designed to assess the effectiveness of the AI system in identifying individuals at risk for BDD, facilitating timely psychological interventions, and improving surgical outcomes.

Study Overview:

Study Population and Inclusion Criteria: Patients aged 18 and older seeking elective cosmetic surgery at a solo practice are included. All participants complete a comprehensive AI-based risk assessment, which includes the Body Dysmorphic Disorder Questionnaire (BDDQ) integrated within the AI system.

AI-Based Risk Assessment: The AI system utilizes data from the BDDQ, along with demographic and psychological factors, to generate a risk score for BDD. This risk score informs the clinical decision-making process, particularly in determining the eligibility for surgery and the need for psychological intervention.

Data Collection and Management: Data is collected through a secure online platform where participants complete the necessary questionnaires. The AI system analyzes the data to generate individualized risk profiles. The study implements rigorous quality assurance processes, including automated data validation checks and source data verification, to ensure the reliability and accuracy of the data.

Statistical Analysis: The study employs correlation analysis to explore the relationships between BDD, age, gender, and stress levels. Chi-square tests are used to assess the statistical significance of differences between demographic groups. The analysis plan includes handling missing data through imputation techniques and conducting sensitivity analyses to validate the robustness of the findings.

Outcome Measures: Primary outcomes include the prevalence of BDD among the study population and the correlations between BDD and key demographic factors. Secondary outcomes focus on the effectiveness of the AI system in enhancing surgical decision-making and improving patient satisfaction.

Ethical Considerations: The study adheres to ethical guidelines, including obtaining informed consent from all participants and anonymizing data to protect privacy. The study is conducted in accordance with the Declaration of Helsinki, and institutional review board approval was deemed unnecessary due to the non-invasive nature of the screening.

Study Limitations: The study acknowledges potential limitations, including the relatively small number of patients who proceeded with surgery, which may affect the generalizability of the findings. Further research is recommended to explore the AI system's effectiveness across diverse populations and clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Completion of the AI-based Body Dysmorphic Disorder Questionnaire (BDDQ)

Exclusion Criteria:

* Individuals under the age of 18 years
* Incomplete or refusal to complete the BDDQ

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes individuals aged 18 years or older who are seeking elective cosmetic surgery at a private practice in Buenos Aires, Argentina. All participants are required to complete an AI-based Body Dysmorphic Disorder (BDD) screening questionnaire as part of the preoperative evaluation. The study aims to assess the prevalence of BDD and its correlation with various risk factors within this population.
Sampling Method: Probability Sample
Enrollment: 3722 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Prevalence of Body Dysmorphic Disorder (BDD) Among Cosmetic Surgery Patients | From 1 to 43 months post-surgery (January 2021 to August 2024)
  This outcome measure assesses the prevalence of BDD among patients undergoing cosmetic surgery, as identified through the AI-powered screening tool.

SECONDARY OUTCOMES:
Correlation Between Positive BDD Screening and Risk Factors | From 1 to 43 months post-surgery (January 2021 to August 2024)
  This measure evaluates the correlation between a positive Body Dysmorphic Disorder (BDD) screening result and various risk factors, including demographic factors (age, gender), psychological stress levels, and previous psychiatric history. The goal is to identify patterns that could inform better patient selection and management in cosmetic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Williams E Bukret, MD, EMBA, Principal Investigator — Bukret Plastic Surgery
Locations (1):
- Bukret Plastic Surgery, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study will be shared after de-identification. Data will be available to other researchers upon reasonable request, subject to approval by the principal investigator, Dr. Williams Erik Bukret. The data will be shared through a secure data-sharing platform.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting information will be available starting 6 months after publication of the study results and will remain available for 1 year.
Access Criteria: IPD and supporting information will be available to researchers who provide a methodologically sound proposal, which must be approved by the principal investigator, Dr. Williams Erik Bukret. Access will be granted for the purpose of academic research, and the data will be shared through a secure data-sharing platform upon request.
URL: https://drbukret.com/research-ipd-sharing/

REFERENCES:
- [Result] Singh AR, Veale D. Understanding and treating body dysmorphic disorder. Indian J Psychiatry. 2019 Jan;61(Suppl 1):S131-S135. doi: 10.4103/psychiatry.IndianJPsychiatry_528_18. PMID 30745686
- [Result] Jabeen M, Shahzadi M, Hussain A, Unbrin A, Ehsaan S. Evaluating internet-based Cognitive Behavioural Therapy (CBT) for body dysmorphic disorder: A systematic review. J Pak Med Assoc. 2024 Aug;74(8):1488-1494. doi: 10.47391/JPMA.10974. PMID 39160718
- [Result] McGrath LR, Oey L, McDonald S, Berle D, Wootton BM. Prevalence of body dysmorphic disorder: A systematic review and meta-analysis. Body Image. 2023 Sep;46:202-211. doi: 10.1016/j.bodyim.2023.06.008. Epub 2023 Jun 21. PMID 37352787
- [Result] Panayi A. The Prevalence of Body Dysmorphic Disorder in Patients Undergoing Cosmetic Surgery: a Systematic Review. Psychiatr Danub. 2015 Sep;27 Suppl 1:S438-44. PMID 26417812
- [Result] Phillipou A, Rossell SL, Wilding HE, Castle DJ. Randomised controlled trials of psychological & pharmacological treatments for body dysmorphic disorder: A systematic review. Psychiatry Res. 2016 Nov 30;245:179-185. doi: 10.1016/j.psychres.2016.05.062. Epub 2016 Aug 5. PMID 27544783
- [Result] Bukret WE. A Novel Artificial Intelligence-assisted Risk Assessment Model for Preventing Complications in Esthetic Surgery. Plast Reconstr Surg Glob Open. 2021 Jul 27;9(7):e3698. doi: 10.1097/GOX.0000000000003698. eCollection 2021 Jul. PMID 34422520
- [Result] Veale D, Gledhill LJ, Christodoulou P, Hodsoll J. Body dysmorphic disorder in different settings: A systematic review and estimated weighted prevalence. Body Image. 2016 Sep;18:168-86. doi: 10.1016/j.bodyim.2016.07.003. Epub 2016 Aug 4. PMID 27498379

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT06584305/Prot_SAP_000.pdf